CLINICAL TRIAL: NCT00252304
Title: Efficacy of Zinc as Adjuvant Therapy in the Treatment of Severe Pneumonia in Nepalese Children at the Kanti Children's Hospital
Brief Title: Therapeutic Zinc in Childhood Pneumonia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre For International Health (Other)
Collaborators: Tribhuvan University, Nepal (Other); Statens Serum Institut (Other); All India Institute of Medical Sciences (Other); Institut de Recherche pour le Developpement (Other Government); Society for Applied Studies (Other)
Responsible Party: Tor A Strand/ Researcher, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCO-CT-2004-003740-2
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Pneumonia
Keywords: Child, severe pneumonia, Zinc, Nepal, therapeutic
MeSH Terms: conditions — Pneumonia | interventions — Zinc; Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc (Experimental): Zinc sulphate 10 or 20 mg per day
  Interventions: Drug: Zinc (zinc sulphate)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc (zinc sulphate) — Dissolvable zinc tablet 10 mg elemental zinc per day for infants 20 mg elemental zinc per day for children 12 to 35 months
  Other Names: Produced by Nutriset; Malaunay, France
  Arms: Zinc
Drug: Placebo — Placebo
  Other Names: Produced by Nutriset; Malaunay, France
  Arms: Placebo

SUMMARY:
The aim of this study is to assess whether zinc given as adjuvant therapy to standard antibiotic treatment in children hospitalized for severe pneumonia reduces the duration of the severe illness and risk of treatment failure. A randomized double blind placebo controlled clinical trial will be conducted at the Kanti Hospital.

DETAILED DESCRIPTION:
Nepal has an under-five mortality rate of 91/1000 live births. Pneumonia, one of the major killers accounts for the death of 25,000 - 35,000 Nepalese children every year. It is estimated that, on an average, of 1000 children <5 years of age that visit health facilities, 90 have pneumonia of which 4.2 have severe pneumonia. At the Kanti Children's Hospital, respiratory diseases are the most frequent reason for admission and the second most frequent cause of child death Zinc, an important micronutrient, is crucial for the normal function of the immune system as well as the integrity of the respiratory epithelium. Zinc deficiency is associated with an increased incidence and severity of diarrhea and respiratory tract infections. The preventive effect of zinc on diarrheal and respiratory illness has been well documented.

Early in an infection zinc is shifted into the liver from the plasma, bone, skin and intestines. For a child with initial low zinc levels, even relatively trivial infections may cause entry into the vicious cycle of reduced plasma zinc and increased infection severity. Administration of zinc during the acute illness may help in reducing the severity of illness.

The therapeutic effect of zinc in acute diarrhea has been well documented. In a study conducted at Bhaktapur, Nepal, in children 6 to 36 months of age, supplementation with zinc was found to be highly effective in the treatment of acute diarrhea.

The Kanti Children's Hospital in Kathmandu serves as a general and referral hospital for children from all parts of the country. Approximately 25% of all admissions to this hospital are due to pneumonia. Being the only well recognized children's hospital, there is always a constraint for available beds for children presenting with pneumonia. Zinc as an adjuvant to standard treatment of pneumonia with antimicrobials was found to hasten recovery from severe pneumonia in children less than 2 years of age in Bangladesh . If we were to conduct a similar study and prove that zinc does in fact help to shorten the duration of illness in children with severe pneumonia, it would go a long way in contributing to improve case management.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2- 35 months with a history of cough (duration <14days) and difficult breathing of </= 72hours' duration, with lower chest indrawing.
* Availability of informed consent.

Exclusion Criteria:

* Children with severe wasting (<70% NCHS median weight for height)
* Severe anemia (hemoglobin <7 gm/dl.)
* Presence of heart disease with or without signs of cardiac failure.
* Child with a chronic cough (lasting for ≥14 days)
* Documented tuberculosis with ongoing treatment.
* Associated other severe diseases that require special care or surgical intervention.
* Children with concomitant diarrhea with some/severe dehydration
* Children with a history of recurrent wheezing
* Children enrolled in the study within the last 6 months of this visit

Ages: 2 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 641 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Time to cessation of severe pneumonia | Within 2 weeks after enrollment
The period starting from enrolment to the beginning of a 24-hour consecutive period of absence of lower chest indrawing, of hypoxia and of any danger signs. | Recovery from pneumonia within 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sudha Basnet, MD, Principal Investigator — Department of Child Health, Institute of Medicine, Tribhuwan University, Katmandu, Nepal; Tor A Strand, MD, PhD, Study Director — Centre For International Health; Halvor Sommerfelt, MD, PhD, Study Chair — Centre For International Health; Nita Bhandari, MBBS, PhD, Study Chair — Centre For International Health; Prakash S Shrestha, MD, Study Director — Child Health Research Project, Department of Child Health, Institute of Medicine, Maharajganj:; Ramesh K Adhikari, MD, Study Chair — Child Health Research Project, Department of Child Health, Institute of Medicine, Maharajganj:
Locations (1):
- Kanti Children Hospital, Kathmandu, Nepal

REFERENCES:
- [Background] Nepal Demographic and Health Survey, 2001
- [Background] Nepal Ministry of Health, Department of Health Services Annual Report 2000- 2001, Kathmandu
- [Background] Shankar AH, Prasad AS. Zinc and immune function: the biological basis of altered resistance to infection. Am J Clin Nutr. 1998 Aug;68(2 Suppl):447S-463S. doi: 10.1093/ajcn/68.2.447S. PMID 9701160
- [Background] Bahl R, Bhandari N, Hambidge KM, Bhan MK. Plasma zinc as a predictor of diarrheal and respiratory morbidity in children in an urban slum setting. Am J Clin Nutr. 1998 Aug;68(2 Suppl):414S-417S. doi: 10.1093/ajcn/68.2.414S. PMID 9701154
- [Background] Bhutta ZA, Black RE, Brown KH, Gardner JM, Gore S, Hidayat A, Khatun F, Martorell R, Ninh NX, Penny ME, Rosado JL, Roy SK, Ruel M, Sazawal S, Shankar A. Prevention of diarrhea and pneumonia by zinc supplementation in children in developing countries: pooled analysis of randomized controlled trials. Zinc Investigators' Collaborative Group. J Pediatr. 1999 Dec;135(6):689-97. doi: 10.1016/s0022-3476(99)70086-7. PMID 10586170
- [Background] Bhandari N, Bahl R, Taneja S, Strand T, Molbak K, Ulvik RJ, Sommerfelt H, Bhan MK. Substantial reduction in severe diarrheal morbidity by daily zinc supplementation in young north Indian children. Pediatrics. 2002 Jun;109(6):e86. doi: 10.1542/peds.109.6.e86. PMID 12042580
- [Background] Brown KH. Effect of infections on plasma zinc concentration and implications for zinc status assessment in low-income countries. Am J Clin Nutr. 1998 Aug;68(2 Suppl):425S-429S. doi: 10.1093/ajcn/68.2.425S. PMID 9701156
- [Background] Beisel WR. Zinc metabolism in infection. In: Brewer GJ, Prasad AS, eds. Zinc metabolism: current aspects in health and disease. New York: Alan R Liss, 1977: 973-977
- [Background] Cousins RJ, Leinart AS. Tissue-specific regulation of zinc metabolism and metallothionein genes by interleukin 1. FASEB J. 1988 Oct;2(13):2884-90. doi: 10.1096/fasebj.2.13.2458983.
- [Background] Strand TA, Hollingshead SK, Julshamn K, Briles DE, Blomberg B, Sommerfelt H. Effects of zinc deficiency and pneumococcal surface protein a immunization on zinc status and the risk of severe infection in mice. Infect Immun. 2003 Apr;71(4):2009-13. doi: 10.1128/IAI.71.4.2009-2013.2003. PMID 12654820
- [Background] Bhutta ZA, Bird SM, Black RE, Brown KH, Gardner JM, Hidayat A, Khatun F, Martorell R, Ninh NX, Penny ME, Rosado JL, Roy SK, Ruel M, Sazawal S, Shankar A. Therapeutic effects of oral zinc in acute and persistent diarrhea in children in developing countries: pooled analysis of randomized controlled trials. Am J Clin Nutr. 2000 Dec;72(6):1516-22. doi: 10.1093/ajcn/72.6.1516. PMID 11101480
- [Background] Strand TA, Chandyo RK, Bahl R, Sharma PR, Adhikari RK, Bhandari N, Ulvik RJ, Molbak K, Bhan MK, Sommerfelt H. Effectiveness and efficacy of zinc for the treatment of acute diarrhea in young children. Pediatrics. 2002 May;109(5):898-903. doi: 10.1542/peds.109.5.898. PMID 11986453
- [Background] Brooks WA, Yunus M, Santosham M, Wahed MA, Nahar K, Yeasmin S, Black RE. Zinc for severe pneumonia in very young children: double-blind placebo-controlled trial. Lancet. 2004 May 22;363(9422):1683-8. doi: 10.1016/S0140-6736(04)16252-1. PMID 15158629
- [Derived] Haugen J, Basnet S, Hardang IM, Sharma A, Mathisen M, Shrestha P, Valentiner-Branth P, Strand TA. Vitamin D status is associated with treatment failure and duration of illness in Nepalese children with severe pneumonia. Pediatr Res. 2017 Dec;82(6):986-993. doi: 10.1038/pr.2017.71. Epub 2017 Aug 16. PMID 28678771
- [Derived] Basnet S, Shrestha PS, Sharma A, Mathisen M, Prasai R, Bhandari N, Adhikari RK, Sommerfelt H, Valentiner-Branth P, Strand TA; Zinc Severe Pneumonia Study Group. A randomized controlled trial of zinc as adjuvant therapy for severe pneumonia in young children. Pediatrics. 2012 Apr;129(4):701-8. doi: 10.1542/peds.2010-3091. Epub 2012 Mar 5. PMID 22392179